CLINICAL TRIAL: NCT00622895
Title: Allogeneic Hematopoietic Cell Transplantation After Nonmyeloablative Conditioning for Patients With Severe Systemic Sclerosis
Brief Title: Allogeneic Hematopoietic Cell Transplantation for Severe Systemic Sclerosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, George Georges, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2067.00; NCI-2011-01352 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R01AI041721 (NIH)
Record Dates: First submitted 2008-02-22; First posted 2008-02-25 (Estimated); Results first posted 2018-06-04 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Systemic Scleroderma; Severe Systemic Sclerosis
Keywords: scleroderma; systemic sclerosis
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse | interventions — fludarabine phosphate; Mycophenolic Acid; Tacrolimus; Whole-Body Irradiation; Bone Marrow Transplantation; Stem Cell Transplantation; Transplantation; Flow Cytometry; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment: allogeneic UCB after reduced intensity conditioning (Experimental): Patients receive fludarabine phosphate IV on days -4, -3 and -2, cyclophosphamide IV over 1-2 hours on days -6, -5, 3, and 4, and undergo low-dose TBI on day -1. Patients receive hematopoietic cell transplantation on day 0.
  Interventions: Drug: fludarabine phosphate; Drug: Mycophenolic Acid; Drug: tacrolimus; Radiation: total-body irradiation; Procedure: bone marrow transplantation; Procedure: reduced intensity allogeneic hematopoietic stem cell transplantation; Procedure: quality-of-life assessment; Other: laboratory biomarker analysis; Other: flow cytometry; Procedure: biopsy

INTERVENTIONS:
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Drug: Mycophenolic Acid — Given PO
  Other Names: Myfortic
Drug: tacrolimus — Given PO
  Other Names: FK 506; Prograf
Radiation: total-body irradiation — Undergo TBI
  Other Names: TBI
Procedure: bone marrow transplantation — Undergo transplantation
  Other Names: stem cell transplantation; progenitor cell transplantation; transplantation
Procedure: reduced intensity allogeneic hematopoietic stem cell transplantation — Undergo transplantation
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: laboratory biomarker analysis — Correlative studies
Other: flow cytometry — Correlative studies
Procedure: biopsy — Punch biopsy of skin involved with scleroderma
  Other Names: biopsies

SUMMARY:
The purpose of the study is to examine the safety and effectiveness of a reduced intensity conditioning regimen and allogeneic bone marrow transplant for people with systemic sclerosis. In an allogeneic bone marrow transplant procedure, bone marrow is taken from a healthy donor and transplanted into the patient. Bone marrow can be donated by a family member or an unrelated donor who is a complete tissue type match.

Participants will receive the chemotherapy and low dose radiation conditioning regimen consisting of the following: Fludarabine will be given intravenously for 5 days. Cyclophosphamide will be given intravenously on the first and second day. After completing the fludarabine and cyclophosphamide, patients will receive a single low dose of total body irradiation. The next day, patients will receive the allogeneic bone marrow transplant. On the third and fourth day after the transplant, patients will receive high dose intravenous cyclophosphamide. This is given to help prevent two complications: (1) graft rejection, which occurs when the body's immune system rejects the donor bone marrow, and (2) graft-versus-host disease (GVHD), which is when the donor immune cells attack the patient's normal tissues. On the fifth day after the transplant, patients will start receiving two additional medications: tacrolimus and mycophenolic acid (MPA, Myfortic), to help prevent GVHD. Patients will receive mycophenolic acid for about 5 weeks and tacrolimus for about 6 months. Also beginning on the fifth day after the transplant, patients will receive daily injections of a growth factor called granulocyte-colony stimulating factor (G-CSF), which is a protein that increases the white blood cell count; G-CSF will be continued until the patient's white blood cell count has returned to normal levels.

Patients will remain closely monitored either in the outpatient clinic setting or in the hospital for approximately 2-3 months after the transplant, but possibly longer if there are complications. Follow-up study visits will occur at 6 months and then at 1, 2, 3, 4, and 5 years after the transplant. Study researchers will keep track of the patient's medical condition after leaving the transplant center by phone calls or mailings to patients and their doctors once a year for the rest of the study participants' lives.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and potential efficacy of reduced intensity conditioning with fludarabine/cyclophosphamide/low-dose total body irradiation (TBI) and allogeneic hematopoietic cell transplantation (HCT) for the stabilization or regression of disease manifestations of severe systemic sclerosis (SSc).

SECONDARY OBJECTIVES:

I. To determine whether stable allogeneic donor engraftment can be safely established with reduced intensity conditioning followed by matched sibling or unrelated donor bone marrow transplantation in patients with severe SSc.

OUTLINE:

Patients receive fludarabine phosphate intravenously (IV) on days -6, -5, -4, -3 and -2 and Cyclophosphamide IV on days -6, -5, and undergo 2 Gray TBI on day -1. Patients receive human leukocyte antigen (HLA)-matched donor bone marrow transplantation on day 0. Patients then receive cyclophosphamide IV on days +3 and +4, and beginning day +5 they start tacrolimus orally (PO) and enteric coated mycophenolic acid.

After completion of initial study treatment, patients are followed up at 6 months and then annually for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for the study must have a human leukocyte antigen (HLA)-identical sibling or HLA-matched unrelated bone marrow donor available and willing to donate.
* Patients with severe SSc as defined by the American College of Rheumatology and at high-risk for a fatal outcome based on the following prognostic factors in groups 1-5:
* Group 1: Patients must have 1) both a and b below; and 2) at least one of c, d or e:

  * a. diffuse cutaneous scleroderma with skin score of greater than or equal to 16 (modified Rodnan scale [mRSS]).
  * b. duration of systemic sclerosis less than or equal to 7 years from the onset of first non-Raynaud's symptom.
  * c. presence of interstitial lung disease (either forced vital capacity [FVC] or corrected diffusing capacity of the lung for carbon monoxide [DLCOcorr] less than 70 % of predicted) and evidence of alveolitis (abnormal bronchoalveolar lavage (BAL) or high resolution chest computed tomography [CT] scan) after treatment with intravenous cyclophosphamide greater than or equal 2 grams given over at least a 3 month period; for patients not able to adequately complete pulmonary function tests (PFT), there must be evidence of progressive disease on chest CT.
  * d. left heart failure with left ventricular ejection fraction (LVEF) < 50% (that has responded to treatment targeted to scleroderma); 2nd or 3rd atrioventricular (AV) block with other evidence of cardiomyopathy related to SSc; myocardial disease not secondary to SSc must be excluded by a cardiologist.
  * e. history of SSc-related renal disease that is not active at the time of screening; history of scleroderma hypertensive renal crisis is included in this criterion.
* Group 2: Progressive pulmonary disease as defined by a decrease in the FVC or DLCOcorr by 15 percent or greater compared to a prior FVC or DLCOcorr in the previous twelve month period; in addition, patients may have either less skin involvement than group 1 (mRSS less than 16) and the FVC or DLCOcorr is less than 70% or both FVC and DLCOcorr greater than or equal to 70% if they have diffuse cutaneous disease (mRSS greater than 16) at screening for the study; patients must also have evidence of alveolitis as defined by abnormal chest CT or BAL; for patients not able to adequately complete PFT, there must be evidence of progressive disease on chest CT.
* Group 3: Have progressive active SSc after prior autologous transplant based on the presence of progressive pulmonary disease; this will be defined by a decrease in the FVC or DLCO adjusted since prior autologous transplant of 15 percent or greater of the pre-transplant percent predicted value, in addition to evidence of alveolitis as defined by chest CT changes or BAL. If patients had prior autologous HCT on the "Scleroderma: Cyclophosphamide Or Transplantation" (SCOT) clinical trial, they must have failed based on the defined study endpoints and be approved by the protocol principal investigator (PI).
* Group 4: Patients who meet group 1 inclusion criteria but may have FVC or DLCO-adjusted less than 70% plus have had an adverse event on cyclophosphamide preventing its further use (specifically hemorrhagic cystitis, leukopenia with white blood cell [WBC]< 2000 or absolute neutrophil count [ANC] < 1000 or platelet count < 100,000).
* Group 5: Diffuse scleroderma with disease duration less than or equal to 2 years since development of first sign of skin thickening plus modified Rodnan skin score greater than or equal to 25 plus erythrocyte sedimentation rate (ESR) > 25 mm/1st hour and/or hemoglobin (Hb) < 11 g/dL, not explained by causes other than active scleroderma.
* Unless patients have a DLCO-adjusted less than 45%, patients in all groups must have failed either oral or intravenous cyclophosphamide regimen defined as: IV cyclophosphamide administration for at least > 3 months between first and last cyclophosphamide dose at a total cumulative IV dose of at least 2 grams, oral cyclophosphamide administration for > 4 months regardless of dose, or combination of oral and IV cyclophosphamide for at least > 6 months independent of dose.
* DONOR: HLA genotypically identical sibling or unrelated donor; unrelated donors are required to be matched by standard molecular methods at the intermediate resolution level at HLA-A, B, C and DRB1 and the allele level at DQB1.
* DONOR: Donors must meet the selection criteria as defined by the Foundation for the Accreditation of Cell Therapy (FACT) and will be screened per the American Association of Blood Banks (AABB) guidelines
* DONOR: Bone marrow is the preferred cell source

Exclusion Criteria:

* Fertile men or women unwilling to use contraceptive techniques during and for 12 months following transplant
* Evidence of ongoing active infection
* Pregnancy
* Patients with a creatinine clearance < 60 ml/min/1.73 m^2 body surface area
* Uncontrolled clinically significant arrhythmias
* Clinical evidence of significant congestive heart failure (CHF) (New York Heart Association [NYHA] Class III or IV)
* LVEF < 45% by echocardiogram
* Severe pulmonary dysfunction with a hemoglobin corrected DLCO < 30% or FVC < 40% of predicted or O2 saturation < 92% at rest without supplemental oxygen
* Significant uncontrolled pulmonary hypertension defined as: Pulmonary artery peak systolic pressure > 55 mmHg by echocardiogram, or pulmonary artery peak systolic pressure 45-55 mmHg by echocardiogram and mean pulmonary artery pressure by right heart catheterization exceeding 25 mmHg at rest (or 30 mmHg with exercise); or NYHA/World Health Organization (WHO), Class III or IV
* Active hepatitis or liver biopsy evidence of cirrhosis or periportal fibrosis; liver function tests: total bilirubin > 2 x the upper limit of normal and/or serum glutamic pyruvate transaminase (SGPT) and SGPT > 4 x the upper limit of normal
* Patients with poorly controlled hypertension
* Patients whose life expectancy is severely limited by illness other than autoimmune disease
* Patients with poorly controlled bleeding from gastric antral vascular ectasia (GAVE) or other gastrointestinal (GI) sites
* Untreated psychiatric illness, drug/alcohol abuse
* Inability to give voluntary informed consent or guardian's informed consent
* Demonstrated lack of compliance with prior medical care
* Malignancy within the 2 years prior to treatment, excluding adequately treated squamous cell skin cancer, basal cell carcinoma, and carcinoma in situ; treatment must have been completed (with the exception of hormonal therapy for breast cancer) with cure/remission status verified for at least 2 years at time of treatment
* Human immunodeficiency virus (HIV) seropositivity
* DONOR: Identical twin
* DONOR: Current pregnancy
* DONOR: HIV seropositivity
* DONOR: Deemed medically unable to undergo bone marrow harvesting
* DONOR: Current serious systemic illness including uncontrolled infections
* DONOR: Failure to meet institutional criteria for donation as described in the Standard Practice Guidelines

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2006-09-01 (Actual); Primary Completion 2011-11-01 (Actual); Study Completion 2017-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Georges, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (2):
- United States (2):
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Allogeneic HCT After Reduced Intensity Conditioning: Conditioning regimen
  * Day -6: cyclophosphamide 50mg/kg. MESNA will be given for bladder prophylaxis .
  * Day -6, -5, -4: Horse ATG 30mg/kg IV x 3 days.
  * Days -6, -5, -4, -3 and -2: Fludarabine 40 mg/m2/day IV over one hour x 5 days.
  * Day -1: TBI 200 cGy at 6-7 cGy/min from a linear accelerator TBI.
  * Day 0: UCB infusion ( 2 units)
  Day -3: Commence tacrolimus at 0.03 mg/kg/day continuous IV infusion until the patient is tolerating oral intake then convert to oral PO b.i.d., continue to day +180 and taper to day +365.
  Day 0: After UCB transplant on day 0, mycophenolate mofetil will be given 1gm IV t.i.d. until the patient is tolerating oral intake and can convert to 1 gram PO T.I.D. Stop MMF at Day +30, if no acute GVHD, until day +100, and then taper 11% week over 8 weeks.
Period: Overall Study
Arm/Group | Treatment: Allogeneic HCT After Reduced Intensity Conditioning
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients are evaluated pre-transplant for assessment of eligibility criteria including chest CT, pulmonary function tests, echocardiogram, bone marrow biopsy, and physical examination as well as standard pre-transplant infectious disease markers.
Arm/Group | Treatment: Allogeneic HCT After Reduced Intensity Conditioning
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 44 [21 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival (EFS)
Description: The events will be defined as any one of the following: death; respiratory failure; renal failure, as defined by chronic dialysis > or = 6 months or kidney transplantation; occurrence of cardiomyopathy, confirmed by clinical CHF (New York Class III or IV) or LVEF < 30% by echocardiogram, sustained for at least 3 months despite therapy; organ dysfunction specific events must be documented on at least two occasions > or = 3 months apart, or sustained for a 3-month period (documented from the first occurrence).
Time Frame: 2 years
Population: UCB transplant recipients
Measure: Count of Participants; unit: Participants
Groups:
- Treatment: Allogeneic HCT After Reduced Intensity Conditioning: Patients receive fludarabine phosphate IV on days -4, -3 and -2, cyclophosphamide IV over 1-2 hours on days -6, -5, 3, and 4, and undergo low-dose TBI on day -1. Patients receive bone marrow transplantation on day 0. Patients then receive cyclophosphamide IV on days +3 and +4, and beginning day +5 they start tacrolimus orally (PO) and mycophenolic acid.
  fludarabine phosphate: Given IV
  Mycophenolic Acid: Given PO
  tacrolimus: Given PO
  total-body irradiation: Undergo TBI
  bone marrow transplantation: Undergo transplantation
  reduced intensity allogeneic hematopoietic stem cell transplantation: Undergo transplantation
  quality-of-life assessment: Ancillary studies
  laboratory biomarker analysis: Correlative studies
  flow cytometry: Correlative studies
  biopsy: Punch biopsy of skin involved with scleroderma
  cyclophosphamide: Given IV
Arm/Group | Treatment: Allogeneic HCT After Reduced Intensity Conditioning
Number analyzed (Participants) | 3
Participants | 1

2. Secondary Outcome: EFS
Description: event-free survival after umbilical cord blood transplant
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment: Allogeneic UCB After Reduced Intensity Conditioning
Number analyzed (Participants) | 3
Participants | 1

3. Secondary Outcome: Overall Survival
Description: Event is defined as death due to any cause.
Time Frame: Up to 5 years
Population: survival of patients after UCB
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment: Allogeneic HCT After Reduced Intensity Conditioning
Number analyzed (Participants) | 3
Participants | 1

4. Secondary Outcome: Treatment-related Mortality
Description: Defined as death occurring at any time after start of allogeneic HCT and definitely or probably resulting from treatment given in the study and not associated with disease progression.
Time Frame: From time of transplant to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment: Allogeneic HCT After Reduced Intensity Conditioning
Number analyzed (Participants) | 3
Participants | 2

5. Secondary Outcome: Regimen-related Toxicity (Greater Than or Equal to Grade III) as Assessed by Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0
Description: Grades 3, 4 and 5 adverse events will be tracked from the start of mobilization or conditioning until day +100 after transplant or until patient departure from the center, whichever occurs first.
  Certain adverse events are usual and expected after transplant and will only be reported if they are > Grade 4. Some Grade 4 events that are routinely expected (i.e. pancytopenia) will not be reported.
Time Frame: Up to 5 years
Population: 3 patients received umbilical cord blood (UCB) transplant.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment: Allogeneic HCT After Reduced Intensity Conditioning: Patients receive fludarabine phosphate IV on days -4, -3 and -2, cyclophosphamide IV over 1-2 hours on days -6, -5, 3, and 4, and undergo low-dose TBI on day -1. Patients receive bone marrow transplantation on day 0. Patients then receive cyclophosphamide IV on days +3 and +4, and beginning day +5 they start tacrolimus orally (PO) and mycophenolic acid.
  fludarabine phosphate: Given IV
  Mycophenolic Acid: Given PO
  tacrolimus: Given PO
  total-body irradiation: Undergo TBI
  bone marrow transplantation: Undergo transplantation
  reduced intensity allogeneic hematopoietic stem cell transplantation: Undergo transplantation
  cyclophosphamide: Given IV
Arm/Group | Treatment: Allogeneic HCT After Reduced Intensity Conditioning
Number analyzed (Participants) | 3
Participants
  Renal failure | 1
  Diffuse alveolar hemorrhage | 1
  Pneumonitis | 1

6. Secondary Outcome: The Percent of Participants With Definite and Probable Viral, Fungal, and Bacterial Infections
Description: The percent of participants with definite and probable viral, fungal, and bacterial infections after transplant
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment: Allogeneic HCT After Reduced Intensity Conditioning
Number analyzed (Participants) | 3
Participants | 2

7. Secondary Outcome: Quality of Life as Assessed by the Modified Scleroderma Health Assessment Questionnaire (SHAQ)
Description: The questionnaire includes measure of quality of life and measure of the scale of skin tightness, activity level and function specifically designed for patients with systemic sclerosis
Time Frame: Up to 5 years
Population: One patient completed the pre-transplant and 5 year post transplant SHAQ (scleroderma health assessment questionnaire). Score range from 0 to 3. Minimum score: Score of 0 is excellent health. Maximum score: score of 3 is most severely impaired, poor quality of life.
Measure: Number; unit: units on a scale
Arm/Group | Treatment: Allogeneic HCT After Reduced Intensity Conditioning
Number analyzed (Participants) | 1
units on a scale
  pre-transplant SHAQ | 1.125
  5 year post transplant | 0.125
  pre-transplant Raynaud symptoms | 3
  5 year post transplant Raynaud symptoms | 0.5
  pre-transplant Finger ulcer symptoms | 3
  5 year post-transplant Finger ulcer symptoms | 0
  pre-transplant Overall health symptoms | 2.5
  5 year post-transplant overall health symptoms | 0.2

8. Secondary Outcome: Quality of Life as Assessed by the Medical Outcome Short Form (36) Health Survey Instrument (SF-36)
Description: The Medical Outcome Short Form (36) Health Survey instrument (SF-36) is a general assessment of health quality of life with eight components: physical functioning, role limitations due to physical health, pain index, general health perceptions, vitality, social functioning, role limitations due to emotional problems and Mental Health Index. Each domain is positively scored, indicating that higher scores are associated with positive outcome.
Time Frame: Up to 5 years
Population: Pre-transplant (baseline) evaluation of physical functioning. Score from 0 to100 with 0 perfect health and 100 poor health.
  The pre-transplant (baseline) evaluation was completed by study participant. The participant did not complete the 5 year post transplant evaluation.
  The 5 year post-transplant SF32 form was not completed by the patient.
Measure: Number; unit: units on a scale
Arm/Group | Treatment: Allogeneic HCT After Reduced Intensity Conditioning
Number analyzed (Participants) | 1
units on a scale
  SF-36 pretransplant overall score | 49.3
  pretransplant limitations due to physical health | 50
  pretransplant limitations due to emotional health | 50

9. Secondary Outcome: Skin Score
Description: The skin score measure is a scale: the name of the scale is the modified Rodnan skin score (mRSS). Total score of mRSS is from 0 to 51. Higher values represents worse skin score. Highest value is 51, represents very hidebound tight thick skin. Lowest value is 0, represent normal skin, no tightness.
Time Frame: Up to 5 years post-transplant
Population: One patient was evaluated at baseline and at 5 years post-transplant. Skin score was evaluated using modified Rodnan skin score (mRSS).
Measure: Number; unit: units on a scale (mRSS)
Arm/Group | Treatment: Allogeneic HCT After Reduced Intensity Conditioning
Number analyzed (Participants) | 1
units on a scale (mRSS)
  Pre-transplant (baseline) skin score | 17
  5 year post-transplant skin score | 4

10. Secondary Outcome: Incidence of Graft Rejection
Description: Engraftment is defined as achieving > 5% donor peripheral blood T cell chimerism by Day 56 after HCT. Primary graft failure is defined as a donor peripheral blood T cell chimerism peak of < 5% by Day 56 post-HCT. Methodological requirements for chimerism are as defined by institutional standard of practice. Secondary Graft Failure is defined as documented engraftment followed by loss of the graft with donor peripheral blood T cell chimerism < 5% as demonstrated by a chimerism assay
Time Frame: Up to day +56
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment: Allogeneic HCT After Reduced Intensity Conditioning
Number analyzed (Participants) | 3
Participants | 0

11. Secondary Outcome: Incidence and Severity of Graft-versus-host Disease (GVHD)
Description: The grading of acute and chronic GVHD will follow previously published guidelines and according to institutional standard of practice but will also include capture of symptoms and characterization of alternative causes. The highest level of organ abnormalities, the etiologies contributing to the abnormalities and biopsy results pertaining to GVHD will be identified. Since both GVHD and SSc involve the skin and the gastrointestinal tract, all diagnostic biopsies of these organs will be centrally reviewed by a study pathologist.
Time Frame: Up to 5 years post-transplant
Population: 1 patient out of the 3 patients enrolled was evaluable for both acute and chronic GVHD. The grade of acute GVHD ranges from 0 to 4. Minimum score of 0 is normal or no GVHD. Maximum score of 4 is fatal GVHD.
  Chronic GVHD minimum score is 0 (none), maximum score 3: extensive and severe.
Measure: Number; unit: units on a scale
Arm/Group | Treatment: Allogeneic HCT After Reduced Intensity Conditioning
Number analyzed (Participants) | 1
units on a scale
  acute GVHD severity maximum grade | 2
  chronic GVHD maximum grade | 2

12. Secondary Outcome: Incidence of Disease-modifying Antirheumatic Drugs (DMARDs) Initiated Post Transplant to Modify Disease
Description: Percent of patients treated with DMARDS after allogeneic transplant in order to treat scleroderma disease signs and symptoms.
Time Frame: Up to 5 years post-transplant
Population: 3 patients enrolled were evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment: Allogeneic HCT After Reduced Intensity Conditioning
Number analyzed (Participants) | 3
Participants
  participants requiring DMARDs | 0
  participants evaluable | 3

ADVERSE EVENTS:
Arm/Group | Treatment: Allogeneic HCT After Reduced Intensity Conditioning
All-Cause Mortality (participants affected / at risk) | 2/3
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment: Allogeneic HCT After Reduced Intensity Conditioning (N=3)
Diffuse Alveolar Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Hypoxia
Renal failure (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment: Allogeneic HCT After Reduced Intensity Conditioning (N=3)
GVHD (Skin and subcutaneous tissue disorders) | 1 (3) — Skin graft versus host disease

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No